CLINICAL TRIAL: NCT04592939
Title: Randomized Controlled Trial of Weight Bearing Status Following Femoral Revision With Tapered, Fluted, Titanium Stems
Brief Title: Trial of Weight Bearing Status Following Femoral Revision With Tapered, Fluted, Titanium Stems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMC20D.220
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Postoperative Pain; Hip Arthroplasty
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: immediate weight bearing (Other)
  Interventions: Procedure: immediate weight bearing after surgery
- Group 2: 6 week toe touch weight bearing (Other)
  Interventions: Procedure: 6 weeks of toe-touch weight bearing after surgery

INTERVENTIONS:
Procedure: immediate weight bearing after surgery — immediate weight bearing
  Arms: Group 1: immediate weight bearing
Procedure: 6 weeks of toe-touch weight bearing after surgery — 6 weeks of toe-touch weight bearing
  Arms: Group 2: 6 week toe touch weight bearing

SUMMARY:
This is a prospective, randomized controlled trial of all patients undergoing femoral revision at Thomas Jefferson University Hospital and Rothman Institute undergoing femoral revision surgery with the use of a modern titanium, fluted, tapered stem. At the time of surgery, patients will be randomized to six weeks of toe-touch weight bearing or immediate weight bearing as tolerated

ELIGIBILITY:
Inclusion Criteria:

* femoral revision patients with the use of a modern titanium, fluted, tapered stem.

Exclusion Criteria:

* include cemented fixation of the stem and patients with a tenuous acetabular reconstruction for whom the surgeon would like to protect weight bearing

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2020-10-19 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Return to function | 1 year
  time to return to baseline ambulatory status
Postoperative Complications | 1 year
  radiographic measurements of subsidence of the stem
Implant survival | 1 year
  re-revision rates within one year

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States